CLINICAL TRIAL: NCT03348956
Title: Biomarkers in Chemotherapy-Induced Peripheral Neurotoxicity: Better Tools and Understanding
Brief Title: Biomarkers in Chemotherapy-Induced Peripheral Neurotoxicity
Acronym: CIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Disarm Therapeutics (Industry)
Responsible Party: Principal Investigator, Victoria H. Lawson, Assistant Professor of Neurology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D17062
Record Dates: First submitted 2017-10-19; First posted 2017-11-21 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: CIPN - Chemotherapy-Induced Peripheral Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EPR Oximetry (Experimental): All subjects in the study will receive the paramagnetic India ink injection to the foot. At three time points (pre-exposure, during-exposure or CIPN incidence, and post exposure), subjects will have three EPR oximetry readings, a neurological examination, and electrophysiologic testing.
  Interventions: Diagnostic Test: EPR Oximetry

INTERVENTIONS:
Diagnostic Test: EPR Oximetry — Subjects will have up to five EPR oximetry readings at each study visit. Subjects will place the foot with the paramagnetic ink injection between the two magnets of the EPR device. Continuous scans will be acquired for 10 minutes while the subject breathes room air, 10 minutes while the subject breathes enriched 100% oxygen, and 10 minutes while breathing room air again.

SUMMARY:
This pilot study will attempt to establish the feasibility of using tissue oxygen measurements and the protein, neurofilament light chain (NF-L), as potential biomarkers for chemotherapy-induced peripheral neuropathy (CIPN). Thirty (30) subjects scheduled to begin taxane-based chemotherapy for breast tumor will be assigned to receive an India ink injection under the skin of the foot. The ink will be used to make up to five (5) 45-minute "electron paramagnetic resonance" (EPR) oximetry readings prior to the start of chemotherapy. Subjects will undergo electrophysiologic assessments including nerve conduction studies, in addition to a neurological examination prior to the start of chemotherapy. Subjects will have the EPR oximetry readings, electrophysiologic tests, and neurological examination two more times: at the halfway point of their chemotherapy treatment -- or at the onset of CIPN symptoms -- and again after chemotherapy has been completed. Subjects will also have blood drawn prior to beginning taxane-based chemotherapy, prior to every scheduled chemotherapy treatment, and after completion of chemotherapy in order to test for neurofilament light chain (NF-L).

DETAILED DESCRIPTION:
Therapy with chemotherapeutic drugs can make a huge impact on survival and quality of life in patients with cancer. Advances in medical monitoring and the effectiveness of these therapies have significantly improved outcomes so that a definitive cure or long-term survival is more likely. Cancer survivors are used to dealing with serious side effects of their therapy; however, some of the side effects from the chemotherapy drugs persist even after the medication course is completed. The impact of these sequelae on quality of survival is increasingly being appreciated and forming an important new direction of cancer care. One of the more severe side effects of chemotherapy is peripheral neurotoxicity resulting in neuropathy or neuronopathy.

Chemotherapy-induced peripheral neurotoxicity (CIPN) is one of the least predictable and most prolonged sequelae with effects ranging from pain, numbness and tingling to diffuse weakness sometimes to the extent of paralysis. It results from damage or alteration in function of peripheral nerves usually, but not always, in a length-dependent manner. An indirect impact of CIPN includes difficulties with balance and susceptibility to falls. There are currently no therapies that have been proven to prevent CIPN. Similarly, there are few medications that are known to be effective in the reversing CIPN once it develops or effectively treating symptoms of CIPN. Currently, diagnosis is based mainly on clinical examination and electrophysiological testing to monitor CIPN; identification of candidate biomarkers through which disease onset can be identified at an earlier stage and which reflect presumed pathophysiologic mechanisms is of paramount importance.

There are different theories of CIPN pathogenesis. One of the leading hypotheses relates to mitochondrial dysfunction and oxidative stress affecting both the dorsal root ganglia neurons and supportive endothelial cells of the vasa nervorum. Here at Dartmouth, a specialized technique has been developed that allows the non-invasive assessment of tissue oxygen in and around peripheral nerve. This technique, called "electron paramagnetic resonance" (EPR) oximetry, allows for repeated measurements over time that can be correlated with other metrics of peripheral nerve function. Given its relevance to an important pathophysiologic mechanism of disease, EPR oximetry may provide an early marker of disease onset.

Neurofilament light chain (NF-L) is also emerging as a sensitive blood-based biomarker of axonal degeneration. NF-L is a component of the axonal cytoskeleton that leaks out of degenerating axons. NF-L has been reported to be elevated in plasma or serum in a wide range of neurodegenerative disorders, including CNS disorders such as multiple sclerosis and ALS as well as PNS disorders such as Charcot Marie Tooth and Guillain-Barre syndrome. To date, there are no published reports of elevated blood NF-L levels in patients with CIPN, although it has been reported to increase in rat model of vincristine-induced neuropathy.

In this proposal, the investigators will be testing the hypothesis that these could both be biomarkers of CIPN. It is hoped that the oximetry measurement and blood NF-L levels will (i) reflect the changes that occur on a cellular level and the damaged nerves, (ii) reflect the damage occurring to nerves more sensitively than existing techniques, and (iii) help to better understand the reason the nerves are being damaged. It is also hoped that these will be something that can be used in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive chemotherapy with taxane compounds for the treatment of breast cancer.
* No prior taxane or platinum chemotherapy prior to enrollment.
* Life expectancy greater than or equal to 12 months.
* Able to provide independent informed consent for the study.
* Able to undergo EPR oximetry
* Age 18 years or older

Exclusion Criteria:

* Central nervous system or other impairments that interfere with clinical and electrophysiological assessment.
* Unable to provide independent informed consent.
* Pacemaker or other metallic objects that would be contraindicated for MRI.
* A requirement for supplemental oxygen at baseline, or known, severe chronic obstructive pulmonary disease .
* Previous exposure to neurotoxic chemotherapeutic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria H Lawson, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center in Lebanon, NH, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not intended to be shared with other researchers per the current protocol and informed consent.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EPR Oximetry
Started | 7
Clinical, Electrophysiologic Metrics, and Neuropathy Scales | 7
Completed | 3
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.5 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in % pO2
Description: EPR Oximetry will measure tissue oxygen levels in the injected foot during 10 minutes of breathing room air, 10 minutes while breathing 100% oxygen, and 10 minutes of room air.
Time Frame: Pre-chemotherapy (Baseline), Mid-chemotherapy (approximately 6 - 8 weeks from Baseline), Post-chemotherapy (approximately 2 - 3 weeks after the participant completed chemotherapy or approximately 14 - 18 weeks from Baseline)
Population: 3 patients underwent testing. 1 patient did not undergo the 100% oxygen condition at the End of Chemo, so there is no data for Mid-Point or recovery for that patient. Data was not gathered for the remaining 4 participants.
Measure: Mean (Full Range); unit: change in % oxygenation
Groups:
- Relative % pO2 Change From Baseline While Breathing Room Air; Relative % pO2 Change From Baseline While Breathing 100% Oxygen; Relative % pO2 Change From Baseline While Breathing Room Air (Recovery): All subjects in the study will receive the paramagnetic India ink injection to the foot. At three time points: pre-exposure (Baseline), during-exposure or CIPN incidence (Mid-Point), and post exposure (End of chemo), subjects will have three EPR oximetry readings, a neurological examination, and electrophysiologic testing.
  EPR Oximetry: Subjects will have EPR oximetry readings at each study visit. Subjects will place the foot with the paramagnetic ink injection between the two magnets of the EPR device. Continuous scans will be acquired for 10 minutes while the subject breathes room air, 10 minutes while the subject breathes enriched 100% oxygen, and 10 minutes while breathing room air again.
Arm/Group | Relative % pO2 Change From Baseline While Breathing Room Air | Relative % pO2 Change From Baseline While Breathing 100% Oxygen | Relative % pO2 Change From Baseline While Breathing Room Air (Recovery)
Number analyzed (Participants) | 3 | 3 | 3
change in % oxygenation
  Mid-Point | 12.3 [-7 to 45] | 19 [-25 to 44] | 24 [11 to 44]
  End of Chemo: number analyzed (Participants) | 3 | 2 | 2
  End of Chemo | 25.3 [20 to 32] | 9.5 [4 to 15] | 42.5 [39 to 46]

2. Secondary Outcome: Neurologic Examination_ Strength_ Toe Fan
Description: Patients will be phenotyped by a neurologic examination before and after exposure to a standard regimen of neurotoxic chemotherapy.
  MRC scale for muscle strength (0-5) Grade 5: Normal Grade 4: Movement against gravity and resistance Grade 3: Movement against gravity over (almost) the full range Grade 2: Movement of the limb but not against gravity Grade 1: Visible contraction without movement of the limb (not existent for hip flexion) Grade 0: No visible contraction
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 5 (0)
  Mid | 4.98 (0.06)
  Post | 4.89 (0.27)

3. Secondary Outcome: Neurologic Examination_ Strength_ Toe Flex
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 5 (0)
  Mid | 4.98 (0.06)
  Post | 4.89 (0.31)

4. Secondary Outcome: Neurologic Examination_ Strength_ Inv
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 5 (0)
  Mid | 4.96 (0.09)
  Post | 4.96 (0.09)

5. Secondary Outcome: Neurologic Examination_ Strength_ Ev
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 5 (0)
  Mid | 4.96 (0.09)
  Post | 4.96 (0.09)

6. Secondary Outcome: Neurologic Examination_ Strength_ ADF
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 5 (0)
  Mid | 5 (0)
  Post | 5 (0)

7. Secondary Outcome: Neurologic Examination_ Vibration Sense_Toe
Description: Patients will be phenotyped by a neurologic examination before and after exposure to a standard regimen of neurotoxic chemotherapy.
  The position of the intersect is recorded on an arbitrary scale from 0 to 8 on a Rydel-Seiffer tuning fork once the subject is no longer perceiving vibration.
  The higher the number, the better the vibratory sense.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 6.71 (0.82)
  Mid | 4.66 (3.10)
  Post | 4.53 (2.09)

8. Secondary Outcome: Neurologic Examination_ Vibration Sense_MM
Description: as for outcome 7
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 6.73 (0.80)
  Mid | 6.44 (1.01)
  Post | 5.78 (1.20)

9. Secondary Outcome: Neurologic Examination_ Vibration Sense_Knee
Description: as for outcome 7
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 6.96 (0.86)
  Mid | 7 (0.98)
  Post | 6.10 (0.68)

10. Secondary Outcome: Neurologic Examination_ Vibration Sense_DIP2
Description: as for outcome 7
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 7.82 (0.46)
  Mid | 7.78 (0.57)
  Post | 7.53 (0.66)

11. Secondary Outcome: Neurologic Examination_ Vibration Sense_DIP5
Description: as for outcome 7
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 7.72 (0.61)
  Mid | 7.76 (0.57)
  Post | 7.60 (0.59)

12. Secondary Outcome: Neurologic Examination_ Deep Tendon Reflexes _ Biceps
Description: Patients will be phenotyped by a neurologic examination before and after exposure to a standard regimen of neurotoxic chemotherapy.
  REFLEX SCALE for Deep Tendon Reflexes (DTRs)
  The score ranges from 0 - 9, where 0 is no reflex response (areflexia)/always abnormal, greater than 1 and less than 3 is normal, and 9 is a tap that elicits a repeating reflex (clonus)/always abnormal.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 4.42 (0.51)
  Mid | 3.28 (1.89)
  Post | 2.14 (1.61)

13. Secondary Outcome: Neurologic Examination_ Deep Tendon Reflexes _ Triceps
Description: as for outcome 12
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 4.14 (1.02)
  Mid | 3.14 (1.74)
  Post | 2.57 (1.78)

14. Secondary Outcome: Neurologic Examination_ Deep Tendon Reflexes _ BR
Description: as for outcome 12
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
Units on a scale
  Pre | 4.21 (0.57)
  Mid | 3.28 (1.54)
  Post | 1.92 (1.32)

15. Secondary Outcome: Neurologic Examination_ Deep Tendon Reflexes _ Patella
Description: as for outcome 12
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
units on a scale
  Pre | 4 (0.67)
  Mid | 3.28 (1.13)
  Post | 2.71 (1.63)

16. Secondary Outcome: Neurologic Examination_ Deep Tendon Reflexes _ Achilles
Description: as for outcome 12
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
units on a scale
  Pre | 4.14 (0.77)
  Mid | 1.57 (1.78)
  Post | 1 (1.35)

17. Secondary Outcome: Mean Nerve Conduction Metrics (Amplitude)_DORSAL SURAL
Description: Electrophysiologic testing will measure nerve conduction amplitude in patients before and after exposure to a standard regimen of neurotoxic chemotherapy.
Time Frame: as for outcome 1
Population: Pre- is prior to chemotherapy exposure Mid- is midway through chemotherapy regimen Post- is one week or more after chemotherapy completion
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
uV
  Pre | 6.2 (8.8)
  Mid | 6.3 (7.7)
  Post | 3.5 (4.7)

18. Secondary Outcome: Change in Nerve Conduction Metrics (Amplitude)_MED PLANTAR
Description: as for outcome 17
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
uV
  Pre | 7.5 (7.2)
  Mid | 6.4 (7.1)
  Post | 5.7 (6.9)

19. Secondary Outcome: Change in Nerve Conduction Metrics (Amplitude)_SURAL
Description: as for outcome 17
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
uV
  Pre | 21.9 (13.1)
  Mid | 16.6 (7.0)
  Post | 19.5 (13.4)

20. Secondary Outcome: Mean of the Difference in Nerve Conduction Amplitudes Between Pre-Mid and Pre-Post exposure_Dorsal Sural
Description: Electrophysiologic testing will measure nerve conduction amplitude in patients before and after exposure to a standard regimen of neurotoxic chemotherapy. The outcome measure is reporting the average of the differences in amplitudes Pre-Mid and Pre-Post exposure (for example, the change from Pre and Mid is calculated, and then the change across all participants is averaged).
Time Frame: as for outcome 1
Population: Pre-Mid- is prior to chemotherapy exposure Pre-Post- is one week or more after chemotherapy completion
Measure: Mean (Full Range); unit: uV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
uV
  Pre-Mid-Mean | -0.47 [-2.3 to 1]
  Pre-Post-Mean | -3.87 [-10.7 to 0]

21. Secondary Outcome: Change in Nerve Conduction/Mixed Nerve Amplitudes _Medial Plantar
Description: as for outcome 17
Time Frame: as for outcome 1
Population: Pre-Mid- is prior to chemotherapy exposure Pre-Post- is one week or more after chemotherapy completion
Measure: Mean (Full Range); unit: uV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
uV
  Pre-Mid-Mean | -1.0 [-7.8 to 3.6]
  Pre-Post-Mean | -1.7 [-13.7 to 3.3]

22. Secondary Outcome: Change in Nerve Conduction/Mixed Nerve Amplitudes _Sural
Description: as for outcome 17
Time Frame: as for outcome 1
Population: Pre-Mid- is prior to chemotherapy exposure Pre-Post- is one week or more after chemotherapy completion
Measure: Mean (Full Range); unit: uV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
uV
  Pre-Mid-Mean | -5.2 [-24.3 to 6.5]
  Pre-Post-Mean | -2.3 [-9.5 to 6.7]

23. Secondary Outcome: Change in Nerve Conduction_Motor_ (Amplitude)_Peron-EDB
Description: as for outcome 17
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
mV
  Pre | 4.6 (1.1)
  Mid | 3.4 (1.9)
  Post | 3.4 (2.7)

24. Secondary Outcome: Change in Nerve Conduction_Motor_ (Amplitude)_Peron-TA
Description: as for outcome 17
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
mV
  Pre | 5.2 (1.4)
  Mid | 5.1 (1.3)
  Post | 5.1 (1.9)

25. Secondary Outcome: Change in Nerve Conduction_Motor_ (Amplitude)_Tibial-AH
Description: as for outcome 17
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
mV
  Pre | 9.2 (3.9)
  Mid | 9.0 (5.7)
  Post | 10.1 (6.8)

26. Secondary Outcome: Nerve Conduction Metrics as Measured by Mean Change (Velocity) for Peroneal CMAP AMP, EDB
Description: Electrophysiologic testing will measure nerve conduction velocity in patients before and after exposure to a standard regimen of neurotoxic chemotherapy.
Time Frame: as for outcome 1
Population: For the dorsal sural sensory nerve, a change in mean velocity pre-chemotherapy to mid-chemotherapy is reported as well as the change in mean velocity for pre-chemotherapy to post-chemotherapy
Measure: Mean (Full Range); unit: m/s
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
m/s
  Pre-Mid | -1.1 [-3.9 to 0.5]
  Pre-Post | -1.4 [-4.6 to 0.7]

27. Secondary Outcome: Nerve Conduction Metrics as Measured by Mean Change (Velocity) for Peroneal CMAP, AT
Description: as for outcome 26
Time Frame: as for outcome 1
Population: as for outcome 26
Measure: Mean (Full Range); unit: m/s
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
m/s
  Pre-Mid | 0 [-1.6 to 3.8]
  Pre-Post | 0 [-2.8 to 5.5]

28. Secondary Outcome: Nerve Conduction Metrics as Measured by Mean Change (Velocity) for Tibial CMAP, AH
Description: as for outcome 26
Time Frame: as for outcome 1
Population: as for outcome 26
Measure: Mean (Full Range); unit: m/s
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
m/s
  Pre-Mid | -0.2 [-4.4 to 3.3]
  Pre-Post | 0.9 [-1.6 to 7.3]

29. Secondary Outcome: Nerve Conduction Metrics as Measured by Mean Change (Velocity) for Dorsal Sural CV
Description: as for outcome 26
Time Frame: as for outcome 1
Population: as for outcome 26
Measure: Mean (Full Range); unit: m/s
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
m/s
  Pre-Mid | 1.8 [-4.0 to 13.8]
  Pre-Post | -1.5 [-6.0 to 2.0]

30. Secondary Outcome: Nerve Conduction Metrics as Measured by Mean Change (Velocity) for Med Plantar CV
Description: as for outcome 26
Time Frame: as for outcome 1
Population: For the Med Plantar sensory nerve, a change in mean velocity pre-chemotherapy to mid-chemotherapy is reported as well as the change in mean velocity for pre-chemotherapy to post-chemotherapy
Measure: Mean (Full Range); unit: m/s
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
m/s
  Pre-Mid | -1.2 [-9.6 to 4.3]
  Pre-Post | -3.5 [-18.7 to 3.7]

31. Secondary Outcome: Nerve Conduction Metrics as Measured by Mean Change (Velocity) for Sural CV
Description: as for outcome 26
Time Frame: as for outcome 1
Population: For the Sural sensory nerve, a change in mean velocity pre-chemotherapy to mid-chemotherapy is reported as well as the change in mean velocity for pre-chemotherapy to post-chemotherapy
Measure: Mean (Full Range); unit: m/s
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
m/s
  Pre-Mid | 2.7 [-5.5 to 11]
  Pre-Post | 0.3 [-10.6 to 9.4]

32. Secondary Outcome: Nerve Conduction Metrics as Measured by Mean Change (Velocity) for Peroneal CV, Distal
Description: as for outcome 26
Time Frame: as for outcome 1
Population: For the Peroneal CV, distal sensory nerve, a change in mean velocity pre-chemotherapy to mid-chemotherapy is reported as well as the change in mean velocity for pre-chemotherapy to post-chemotherapy
Measure: Mean (Full Range); unit: m/s
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
m/s
  Pre-Mid | 1.6 [-2.0 to 4.5]
  Pre-Post | -2.2 [-8.3 to 4.1]

33. Secondary Outcome: Mean Score of Neuro-Quality of Life - Positive Affect and Well-Being Scale
Description: Neuropathy-Specific Quality of Life scale measuring Positive Affect and Well Being
  The range in score is 23 to 115, with a low score indicating a less positive affect and well-being
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 93.9 (21.5)
  Mid | 96.3 (17.4)
  Post | 100.6 (17.1)

34. Secondary Outcome: Mean Score of Neuro-Quality of Life - Satisfaction With Social Roles and Activities Scale
Description: Neuropathy-Specific Quality of Life scale measuring Satisfaction with Social Roles and Activities
  The range in scores is 47 to 235, with a lower score indicating less satisfaction with social roles and activities
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 172.9 (46.4)
  Mid | 187.1 (33.5)
  Post | 187.6 (50.0)

35. Secondary Outcome: Mean Score of Neuro-Quality of Life - Lower Extremity Function (Mobility) Scale
Description: Neuropathy-Specific Quality of Life scale measuring Lower Extremity Function (Mobility)
  The range in scores is 19 to 95, with a lower score indicating more difficulty with lower extremity function
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 89.1 (10.1)
  Mid | 90.6 (7.1)
  Post | 91.4 (5.9)

36. Secondary Outcome: Mean Score of Neuro-Quality of Life - Upper Extremity Function (Fine Motor, Activities of Daily Living) Scale
Description: Neuropathy-Specific Quality of Life scale measuring Upper Extremity Function (Fine Motor, Activities of Daily Living)
  The range in scores is 20 to 100, with a low score indicating more difficulty with upper extremity function
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 97.0 (5.5)
  Mid | 99.3 (1.5)
  Post | 97.9 (4.4)

37. Secondary Outcome: Mean Score of The Neuropathy Total Symptom Score-6 Questionnaire
Description: Neuropathy Total Symptom Score questionnaire with 6 questions
  The range is scores is 0 to 22 with a higher score indicating worse symptoms
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 0.3 (0.5)
  Mid | 2.2 (1.8)
  Post | 3.1 (3.1)

38. Secondary Outcome: Mean Score of Toronto Clinical Neuropathy Scoring System
Description: Toronto Clinical Neuropathy Scoring System
  The range in scores is 0 to 19 with higher scores indicating worse neuropathy
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 2.1 (2.0)
  Mid | 5.3 (3.4)
  Post | 5.0 (3.7)

39. Secondary Outcome: Mean Score of National Cancer Institute - Common Toxicity Criteria
Description: National Cancer Insitute - Common Toxicity Criteria
  The range in scores is 0 to 5, with higher scores indicating worse toxicity
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 0.3 (0.8)
  Mid | 0.7 (1.0)
  Post | 1.4 (0.8)

40. Secondary Outcome: Mean Score of Total Neuropathy Scores
Description: Total Neuropathy score
  The range in scores is 0 to 40, with higher scores indicating worse neuropathy
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 1.3 (1.1)
  Mid | 6.0 (5.0)
  Post | 8.1 (6.2)

41. Secondary Outcome: Mean Score of Survey of Autonomic Symptoms, Column B
Description: Survey of Autonomic Symptoms, questions in Column B
  The range in scores is 0 to 55 for women and 0 to 60 for men, with higher scores indicating more bothersome symptoms
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 5.9 (3.7)
  Mid | 6.9 (4.9)
  Post | 5.2 (3.9)

42. Secondary Outcome: Mean Score of McGill Pain Visual Analog Scale
Description: McGill Visual Analog Scale for Pain
  The range in scores is 0 to 100, with 0 indicting "No pain" and 100 indicating "Worst pain possible"
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 21.0 (23.8)
  Mid | 27.9 (25.5)
  Post | 27.3 (30.9)

43. Secondary Outcome: Mean Scores of Short Form McGill Pain Questionnaire
Description: Short Form McGill Pain Questionnaire
  The range in scores is 0 to 15, with higher scores indicating worse pain
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 3.3 (4.0)
  Mid | 2.4 (2.1)
  Post | 2.3 (1.9)

44. Secondary Outcome: Mean Score of Survey of Autonomic Symptoms, Column A
Description: Survey of Autonomic Symptoms, questions in column A
  The range in scores is 0 to 11 for women and 0 to 12 for men, with higher scores indicating more symptoms
Time Frame: as for outcome 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 7
score on a scale
  Pre | 2.4 (1.1)
  Mid | 2.3 (0.8)
  Post | 2.0 (1.4)

45. Secondary Outcome: Serum NF-L Levels
Description: Changes in serum NFL levels over the course of chemotherapy will be monitored to determine if NFL can be used as a biomarker for axonal damage in patients who develop CIPN. NFL will be measured at baseline, before each round of chemotherapy and at the completion of chemotherapy. Changes in NFL will be compared between patients who develop CIPN and those that do not.
Time Frame: 1 year
Population: Samples were never gathered due to no participants enrolled after protocol was amended to include the collection of serum NF-L.
Arm/Group | EPR Oximetry
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be reported from the initiation of any study procedures to the end of the study treatment follow-up. Adverse events were collected from Baseline through 15 - 18 weeks after chemotherapy.
Arm/Group | EPR Oximetry
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPR Oximetry (N=7)
Erythema (Vascular disorders) | 2 (2) — Erythema on chest wall over mastectomy site
Nausea (General disorders) | 3 (3) — Nausea
Increased symptoms of reflux (General disorders) | 1 (1) — increased symptoms of reflux
Abnormal Lab Values (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
High LFT's (General disorders) | 2 (2)
Increased Fatigue (General disorders) | 3 (3)
Soreness in both walls along MRM incision (General disorders) | 1 (1)
CIPN (Nervous system disorders) | 5 (5) — length-dependent, axonal sensory motor neuropathy
Redness/Itchy on scalp (General disorders) | 1 (1) — Little red bumps on scalp that are itchy
Cramping in calves- severe (General disorders) | 1 (1)
Discomfort in anterior aspect of shins (General disorders) | 1 (1)
Decreased Dexterity (General disorders) | 1 (1)
Increased unsteadiness (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Indigestion (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Sore Throat due to Nocturnal Epistaxis (General disorders) | 1 (1)
Alopecia (General disorders) | 3 (3)
Anemia-Mild (General disorders) | 2 (2)
Dysphagia (General disorders) | 2 (2)
High WBC w/o infection (General disorders) | 3 (3)
Thrush on tongue (General disorders) | 1 (1)
Low K+ Lab (General disorders) | 1 (1)
Diverticulitis (General disorders) | 1 (1)
Shortness of breath (General disorders) | 1 (1)
left ankle swelling-occasional (General disorders) | 1 (1)
Pain during urination (General disorders) | 1 (1)
Worsening Appetite (General disorders) | 1 (1)
Knee Pain (General disorders) | 1 (1)
Pain up to hip from knee (General disorders) | 1 (1)
Shingles (General disorders) | 1 (1)
Cellulitis (General disorders) | 1 (1)
Bloating (General disorders) | 1 (1)
Dry Mouth (General disorders) | 1 (1)
Hyperhidrosis (General disorders) | 1 (1)
Brief periods of heart pounding (General disorders) | 1 (1)
Aches, Cramps and Spasms (General disorders) | 1 (1)
Sore on tip of tongue (General disorders) | 1 (1)
Brief burning sensation on chest, back, and legs (General disorders) | 1 (1)
Low grade fever (General disorders) | 1 (1)
Ecchymosis (General disorders) | 1 (1)
Bilateral ankle swelling (General disorders) | 1 (1)
Myalgia (General disorders) | 1 (1)
Cytopenia (General disorders) | 1 (1)
Discomfort at Injection Site (General disorders) | 1 (1)
Right Hip/Lower back pain (General disorders) | 1 (1)
Myalgias (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Mild Cough (General disorders) | 1 (1)
Mild Anemia (General disorders) | 1 (1)
Arthralgias (General disorders) | 1 (1)
Dysgeusia (General disorders) | 1 (1)
Acute Pharyngitis (General disorders) | 1 (1)
Pain at injection site (General disorders) | 1 (1)
Purple Hematoma at injection site (General disorders) | 1 (1)
Rash-under Arm Pit (General disorders) | 1 (1)
Redness along hands and wrists (General disorders) | 1 (1)
Mouth Sore (General disorders) | 1 (1)
Tearing of eyes (General disorders) | 1 (1)
Allergic Reaction (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
LIMITATION OF EPR DATA While it may be feasible to make serial measurements with the technique, there were technical problems with the sensor (India Ink), and no conclusions can be drawn in regard to oxygenation. Additionally, the ERP data are limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03348956/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT03348956/ICF_001.pdf